CLINICAL TRIAL: NCT04261725
Title: Evaluation of the Prevalence of EGFR Mutations in epidermoïd Bronchopulmonary Cancers Diagnosed in Réunion
Brief Title: Prevalence of EGFR Mutations in epidermoïd Bronchopulmonary Cancers in Réunion Island
Acronym: EPIMURE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/CHU/18
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Squamous Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Squamous Cell Lung Cancer: Genetic analysis for searching EGFR mutation
  Interventions: Genetic: EGFR mutation

INTERVENTIONS:
Genetic: EGFR mutation — Searching the EGFR mutation in pulmonary biopsy

SUMMARY:
Lung cancer is the most common cancer in the world with 1.8 million estimated incident cases in 2012 (12.9% of diagnosed cancers) and 1.6 million deaths annually. In mainland France, lung cancer represents 12% of all incident cancers. The standardized incidence rates for the world population were then 52.6 per 100,000 for men and 23.4 / 100,000 for women, respectively. In Reunion, 415 cases of primary bronchopulmonary cancers were reported for the years 2011-2012, which gives standardized incidence rates lower than those observed in mainland France (33.1 / 100,000 in humans, 8.2 / 100,000 in women).

If the incidence of bronchopulmonary cancer is lower in Réunion than in mainland France, the study of histological subtypes appears different: the investigators observe a greater frequency of adenocarcinomas (65% vs 45%), at the expense squamous cell carcinomas. In addition, for adenocarcinomas, the frequency of EGFR type mutations is twice as high (23% vs 11%). Thus, if this rate of EGFR mutations observed in mainland France is very close to those described in all Caucasian populations, that observed in the Reunionese population appears closer to those described in Asian populations, and more particularly the Indian population. This can perhaps be explained by the fact that the population of Reunion is a cosmopolitan and highly mixed race, whose share of Asian origin, mainly Indian and Chinese, is significant.

In clinical practice, INCa recommends carrying out the search for the EGFR mutation for any patient with locally advanced or metastatic lung carcinoma, not small cell and non epidermoid. This restriction to the histology of adenocarcinoma is justified by the low frequency of EGFR mutations for other histological types in Caucasian populations. However, some studies describe significant EGFR mutation rates for epidermoid cancers in Asian populations, particularly in India. Thus, given that a large part of the Réunion population shares Asian origins, the question of the frequency of EGFR mutations among squamous cell carcinomas in Réunion is asked.

The hypothesis of this research is that, given the ethnic characteristics of the Reunionese population, the proportion of bronchopulmonary epidermoid cancers carrying the EGFR mutation is potentially significantly higher than that observed in Caucasian populations, including the French metropolitan population. If this rate of EGFR mutations were high in the Reunion population, it would then be necessary to allow the search for this mutation to be extended to all bronchopulmonary cancers, which will improve their therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over,
* who is diagnosed with bronchopulmonary squamous cell carcinoma in one of the 2 anatomopathology laboratories at Reunion University Hospital,

Exclusion Criteria:

- refuses to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with bronchopulmonary squamous cell carcinoma in one of the 2 anatomopathology laboratories at Reunion University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of EGFR mutations among bronchopulmonary squamous cell carcinomas | 1 month
  Proportion of bronchopulmonary squamous cell carcinomas carrying the EGFR mutation among all bronchopulmonary squamous cell carcinomas treated at the CHU de la Réunion and at the Clinique Sainte Clotilde and whose histological diagnosis was carried out in one of the two laboratories anatomopathology of the University Hospital of Réunion.

CONTACTS AND LOCATIONS:
Overall Officials: Michel ANDRE, MD, Principal Investigator — Centre Hospitalier Universitaire de la Réunion
Locations (3):
- Reunion (3):
  - Centre Hosiptalier Universitaire de La Réunion - site Nord, Saint-Denis
  - Centre Hospitalier niversitaire - site Sud, Saint-Pierre
  - Clinique Saint Clotilde, Sainte-Clotilde

IPD SHARING:
Plan to Share IPD: No